CLINICAL TRIAL: NCT06668909
Title: Patient Reported Outcomes on Vision Quality and Dry Eye Following Treatment With Wavelight LASIK
Brief Title: Patient Reported Outcomes With WaveLight LASIK
Status: Completed | Type: Observational
Sponsor: OVO LASIK + Lens (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: ML-24-01
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: WaveLight® EX500 — Phorcidies Planned Contoura LASIK

SUMMARY:
This study is a multi-site, single-arm, ambispective, observational study of subject satisfaction, after successful bilateral LASIK surgery. Subjects will be assessed 12+ months post-operatively. Clinical evaluations will include administration of the OSDI, modified PROWL, and dry eye questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Wavefront Optimized or Phorcidies Planned Contoura LASIK for myopia or myopic astigmatism 12 to 15 months ago
* Age: 21 to 35 years of age at the time of surgery.
* Preoperative myopic sphere of -1.00 D to -8.00 D
* Preoperative regular astigmatism of 0.00 D to -3.00 D.
* Stable refraction preoperatively defined as < 0.5 D of change over at least 1 year.
* Refractive target of bilateral emmetropia.

Exclusion Criteria:

* Corneal ectatic disorders.
* Patients with a calculated residual stromal depth of < 300 um.
* Pre-existing retinal or corneal pathology, or irregular astigmatism.
* Pre-existing autoimmune diseases, dry eye, glaucoma, diabetes, etc.
* Previous corneal surgeries prior to LASIK.
* LASIK enhancements.

Ages: 21 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Eligible test subjects will be 21 to 35 years of age (at the time of surgery) and who underwent Wavefront Optimized or Phorcidies Planned Contoura LASIK for myopia or myopic astigmatism 12 to 15 months prior.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 12 months postoperatively
  Percentage of subjects satisfied (Completely Satisfied or Very Satisfied) with vision after Wavelight LASIK based on a modified PROWL Questionnaire (Question #1 only).

SECONDARY OUTCOMES:
PROWL Questionnaire | 12 months postoperatively
  PROWL-SS can be used to assess satisfaction with vision and the existence, bothersomeness and impact on usual activities in the last 7 days of four visual symptoms - double images (8 items), glare (8 items), halos (8 items) and starbursts (8 items). Subjects select one of 6 responses for each question.
OSDI Questionnaire | 12 months postoperatively
  The OSDI© is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease. The OSDI© is a valid and reliable instrument for measuring dry eye disease (normal, mild to moderate, and severe) and effect on vision-related function.
Percentage of subjects using artificial tears or prescription dry eye medication. | 12 months postoperatively

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - NVISION Eye Centers, San Diego, California
  - Boston Vision, Brookline, Massachusetts
  - Ovo Lasik + Lens, Saint Louis Park, Minnesota
  - Mann Eye Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No